CLINICAL TRIAL: NCT03950882
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Pharmacokinetics of PXL770 After 4 Weeks of Treatment in Subjects With Non-alcoholic Fatty Liver Disease (NAFLD)
Brief Title: A Study to Assess the Pharmacokinetics of PXL770 After 4 Weeks of Treatment in Subjects With NAFLD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Poxel SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PXL770-003
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Nonalcoholic Fatty Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — 2-chloro-3-(1-hydroxy-5,6,7,8-tetrahydronaphthalen-2-yl)-6-oxo-5-phenyl-7H-thieno)(2,3-b)pyridin-4-olate potassium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PXL770 (Experimental): PXL770 500 mg once daily (QD) for 4 weeks
  Interventions: Drug: PXL770; Drug: Placebo
- Placebo (Placebo Comparator): placebo once daily (QD) for 4 weeks
  Interventions: Drug: PXL770; Drug: Placebo

INTERVENTIONS:
Drug: PXL770 — Oral capsule
Drug: Placebo — Oral capsule

SUMMARY:
This study will assess the pharmacokinetics of PXL770 after 4 weeks of treatment.

DETAILED DESCRIPTION:
The study will be performed in subjects with Nonalcoholic Fatty Liver Disease. The primary endpoint will be the assessment of PXL770 exposure in plasma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have given written informed consent
* Body mass index (BMI): ≥ 25 kg/m²
* Hepatic steatosis (CAP ≥ 300)
* Insulin-resistant but not diabetic subjects
* Fasting plasma glucose <126 mg/dL
* Glomerular filtration rate (eGFR) ≥ 60 mL/[min*1.73 m²]
* Alanine amino transferase (ALT) > 20 IU/L in females and > 30 IU/L in males
* Effective contraception

Exclusion Criteria:

* Evidence of another form of liver disease
* Evidence of liver cirrhosis
* Evidence of hepatic impairment
* Positive serologic evidence of current infectious liver disease
* History of excessive alcohol intake
* Acute cardiovascular disease with 24 weeks prior to screening
* Uncontrolled high blood pressure
* Any disease which in the Investigator's opinion which in the Investigator's opinion would exclude the patient from the study
* Use of non-permitted concomitant medication
* Pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-03-29 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
PK parameters of PXL770 | Day 26
  AUC : Area under the plasma concentration curve

SECONDARY OUTCOMES:
Plasma PK parameters of PXL770 | Day 26
  Minimum plasma concentration (Cmin)
Plasma PK parameters of PXL770 | Day 26
  Average plasma concentration (Cavg)
Plasma PK parameters of PXL770 | Day 26
  Time to maximum plasma concentration (Tmax)
Plasma PK parameters of PXL770 | Day 26
  Apparent volume of distribution (Vz/F)
Plasma PK parameters of PXL770 | Day 26
  Apparent oral drug clearance at steady state (CLss/F)
Plasma PK parameters of PXL770 | Day 26
  Elimination rate constant (λz)
Plasma PK parameters of PXL770 | Day 26
  Terminal elimination half-life (t½)
Plasma PK parameters of PXL770 | Day 26
  Area under the concentration-time curve from time 0 to last observed concentration (AUClast)
Plasma PK parameters of PXL770 | Day 14 and Day 26
  Food effect: Cmax
Plasma PK parameters of PXL770 | Day 14 and Day 26
  Food effect: AUCtau
Plasma PK parameters of PXL770 | Day 14 and Day 26
  Food effect: Tmax
Plasma PK parameters of PXL770 | Day 27
  PK profile during OGTT: AUCtau
Plasma PK parameters of PXL770 | Day 27
  PK profile during OGTT: Cmax

CONTACTS AND LOCATIONS:
Locations (1):
- High Point Clinical Trials Center, High Point, North Carolina, United States

REFERENCES:
- [Derived] Fouqueray P, Bolze S, Dubourg J, Hallakou-Bozec S, Theurey P, Grouin JM, Chevalier C, Gluais-Dagorn P, Moller DE, Cusi K. Pharmacodynamic effects of direct AMP kinase activation in humans with insulin resistance and non-alcoholic fatty liver disease: A phase 1b study. Cell Rep Med. 2021 Dec 21;2(12):100474. doi: 10.1016/j.xcrm.2021.100474. eCollection 2021 Dec 21. PMID 35028615